CLINICAL TRIAL: NCT02282514
Title: Non-myeloablative Hematopoietic Stem Cell Transplantation for Stiff Person Syndrome (SPS) and Anti-GAD Antibody Variants: Progressive Encephalomyelitis With Rigidity and Myoclonus (PERM), and Adult Onset Autoimmune Anti-GAD Positive Cerebellar Ataxia
Brief Title: Stem Cell Transplantation for Stiff Person Syndrome (SPS)
Acronym: SPS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Could not predict who would respond, relapse or go into remission
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, Professor, Division Chief, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIAD.SPS.2014
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Stiff-Person Syndrome
Keywords: Autoimmune Diseases; Autologous Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Stiff-Person Syndrome; Autoimmune Diseases | interventions — Cyclophosphamide; Mesna; thymoglobulin; Methylprednisolone; Methylprednisolone Hemisuccinate; Granulocyte Colony-Stimulating Factor; Filgrastim; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Experimental): The conditioning regimen will be 200 mg/kg of intravenous cyclophosphamide given in 4 equal fractions on days -5 through -2 with intravenous mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5, 1.0 mg/kg on days -4 and -3, and then 1.5 mg/kg on days -2 and -1. Methylprednisolone 1000 mg will be infused intravenously before each dose of rATG. Autologous hematopoietic stem cells will be infused intravenously on day 0. A granulocyte-colony stimulating factor (G-CSF) 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment. Intravenous Rituxan (500mg) will be administered on days -6 and +1.
  Interventions: Biological: Autologous Hematopoietic Stem Cells; Drug: Cyclophosphamide; Drug: Mesna; Drug: rATG; Drug: Methylprednisolone; Drug: G-CSF; Drug: Rituxan

INTERVENTIONS:
Biological: Autologous Hematopoietic Stem Cells — The stem cells will be collected from patient's blood during mobilization. Then the patient will be given high dose chemotherapy in accordance with approved recommendations for use in conditioning regimens for stem cell transplant in autoimmune diseases. Autologous Hematopoietic Stem Cell Transplantation is to re-infuse immature cells that can re-establish blood production and patient's immune system.
Drug: Cyclophosphamide — An alkylating agent which causes prevention of cell division by forming adducts with DNA
  Other Names: Cytoxan; Neosar; Endoxan
Drug: Mesna — Medication used to decrease the risk of hemorrhagic cystitis prophylaxis
  Other Names: Mesnex
Drug: rATG — A predominantly lymphocyte-specific immunosuppressive agent which contains antibodies specific to the antigens commonly found on the surface of T cells
  Other Names: Thymoglobulin
Drug: Methylprednisolone — Steroid
  Other Names: Solu-Medrol
Drug: G-CSF — Granulocyte-colony stimulating factor; a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  Other Names: Neupogen; Filgrastim; Granix; Zarxio
Drug: Rituxan — A chimeric monoclonal antibody used in the treatment of B cell non-Hodgkin's lymphoma, B cell leukemia, and some autoimmune disorders
  Other Names: Rituximab

SUMMARY:
Non-myeloablative regimens (as the investigators use herein) are designed to maximally suppress the immune system without destruction of the bone marrow stem cell compartment.

When using a non-myeloablative regimen recovery occurs without infusion of stem cells and the stem cells are autologous. While not necessary for recovery, stem cell infusion may shorten the interval of neutropenia and attendant complications. Thus in reality there is no transplant only an autologous supportive blood product.

Based on our encouraging results of non-myeloablative hematopoietic stem cell transplantation, for patients with multiple sclerosis and chronic inflammatory demyelinating polyneuropathy, the investigators will investigate the role of non-myeloablative hematopoietic stem cell transplantation for patients with SPS who require assistance to ambulate.

DETAILED DESCRIPTION:
Pre-study Testing

1. History and physical
2. Electrocardiogram (EKG)
3. Dobutamine stress echocardiogram
4. High-resolution computed tomography of the chest (HRCT)
5. Blood draw for laboratory tests- these tests will include a complete blood count, evaluating liver and kidney function, assessing immune system, tissue typing, and checking for certain germs that can cause infections, including a pregnancy test for females and prostate-specific antigen (PSA) for male as well as testing for HIV
6. Pulmonary Function Test (PFT)
7. Electromyography (EMG)
8. Magnetic Resonance Imaging (MRI) of the Abdomen and Pelvis
9. Magnetic Resonance Imaging (MRI) of the Spinal Cord
10. Magnetic Resonance Imaging (MRI) of the Brain with Gadolinium (only if PERM of cerebellar ataxia)
11. Colonoscopy
12. Mammogram (if female)
13. Timed ambulation
14. Quality of Life Questionnaires [ Short Form (36) Health Survey (SF36) and Barthel Index]
15. Chronic Pain Acceptance Questionnaire (CPAQ)
16. Rankin Functional Scale
17. Modified Ashworth Scale
18. Purkinje Cell Cytoplasmic Antibody, Type 1 (PCA-1), Purkinje Cell Cytoplasmic Antibody, Type 2 (PCA-2) antibody (only if cerebellar ataxia)
19. Spinocerebellar ataxia (SCA) 1, 2, 3, 4, 5, 6, 7, 8 genes (only if ataxia)

Study Treatment

Stem Cell Collection: Cyclophosphamide 2.0 gm/m2 will be given on day 0, G-CSF 5-10 mcg/kg/day subcutaneous (SQ) will start on day +5 and will continue until apheresis is discontinued. Apheresis will begin when the absolute neutrophil count (ANC) > 1.0 x 109/L and continue until >2.0 x 106 cluster of differentiation 34 (CD34)+ cells/kg patient weight are cryopreserved. A 10-15 liter apheresis will be performed unless stopped earlier for clinical judgment of toxicity (e.g., numbness, tetany). A maximum of four apheresis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Stiff-person Syndrome and

   * Age between 18 and 60 years old
   * Failure of medically tolerable doses (20-40 mg/day) of diazepam
   * Failure of either intravenous immunoglobulin (IVIg) and or plasmapheresis
   * Stiffness in the axial muscles, prominently in the abdominal and thoracolumbar paraspinal muscle leading to a fixed deformity (hyperlordosis)
   * Superimposed painful spasms precipitated by unexpected noises, emotional stress, tactile stimuli
   * Confirmation of the continuous motor unit activity in agonist and antagonist muscles by electromyography when off diazepam and anti-spasmatic medications
   * Absence of neurological or cognitive impairments that could explain the stiffness
   * Inability to run or walk, or abnormal gait
2. Diagnosis of a SPS variant- Progressive Encephalomyelitis with Rigidity and Myoclonus (PERM) defined as:

   Acute onset of painful rigidity and muscle spasms in the limbs and trunk
   * Brainstem dysfunction (nystagmus, opsoclonus, ophthalmoparesis, deafness, dysarthria, dysphagia)
   * Profound autonomic disturbance.
   * Positive serology for GAD65 (or amphiphysin) autoantibodies, assessed by immunocytochemistry, western blot or radioimmunoassay (>1000 u/ml)
   * MRI may show increased signal intensity throughout the spinal cord and the brainstem
3. Diagnosis of a SPS variant - anti-GAD positive cerebellar ataxia

   * Subacute or chronic onset of cerebellar symptoms-gait or limb ataxia, dysarthria, nystagmus
   * Positive serology for GAD65 (or amphiphysin) autoantibodies, assessed by immunocytochemistry, western blot or radioimmunoassay (>1000 u/ml)
   * Anti-GAD antibody in cerebrospinal fluid
   * Abnormal MRI imaging of brainstem or cerebellum other than cerebellar atrophy
   * Negative history of toxin or alcohol
   * Absence of Vitamin B12 or Vitamin E deficiency
   * Absence of positive HIV, syphilis or whipple disease
   * Absence of consanguinity, positive family history for ataxia or positive genetic screen for spinocerebellar ataxia (SCA) 1, SCA 2, SCA 3, SCA 6, SCA 7 or SCA 8 mutation

Exclusion Criteria:

* Current or prior history of a malignancy or paraneoplastic syndrome
* Inability to sign and understand consent and be compliant with treatment
* Positive pregnancy test
* Inability to or comprehend irreversible sterility as a possible side effect
* Amphiphysin antibody positive
* Left ventricular ejection fraction (LVEF) < 45% or ischemic coronary artery disease on dobutamine stress echocardiogram
* Diffusing capacity of the lungs for carbon monoxide (DLCO) < 60% predicted
* Serum creatinine > 2.0 mg/dl
* Bilirubin >2.0 mg/dl
* Platelet count < 100,000 / ul, white blood cell count (WBC) < 1,500 cells/mm3
* History of toxin or alcohol abuse
* History of Vitamin B12 or Vitamin E deficiency
* Positive HIV, syphilis, or whipple disease
* Consanguinity, positive family history for ataxia or positive genetic screen for SCA1, SCA2, SCA3, SCA6, SCA 7 or SCA8 mutation (if ataxia present)
* Absence of at least one SPS associated antibody such as anti-GAD, or gamma-aminobutyric acid (GABA)-A receptor associated protein, or synaptophysin, or gephyrin, or GABA-transaminase

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-10; Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Burt RK, Balabanov R, Han X, Quigley K, Arnautovic I, Helenowski I, Rose J, Siddique T. Autologous Hematopoietic Stem Cell Transplantation for Stiff-Person Spectrum Disorder: A Clinical Trial. Neurology. 2021 Feb 9;96(6):e817-e830. doi: 10.1212/WNL.0000000000011338. Epub 2020 Dec 14. PMID 33318163

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplantation: Conditioning regimen will be 200 mg/kg of IV cyclophosphamide given in 4 equal fractions on days -5 through -2 with IV mesna. Rabbit antithymocyte globulin (rATG) (Thymoglobulin®) will be dosed at 0.5 mg/kg on day-5, 1.0 mg/kg on days -4 and -3, and then 1.5 mg/kg on days -2 and -1. Methylprednisolone 1000 mg will be infused IV before each dose of rATG. Autologous hematopoietic stem cells (HSCT) will be infused IV on day 0. A granulocyte-colony stimulating factor (G-CSF) 5-10 mcg/kg will be started on day + 5 and continued until neutrophil engraftment. Intravenous Rituxan (500mg) will be administered on days -6 and +1.
  HSCT: cells will be collected from blood during mobilization. Then the patient will be given high dose chemotherapy in accordance with approved recommendations for use in conditioning regimens for stem cell transplant in autoimmune diseases. Autologous HSCT is to re-infuse immature cells that can re-establish blood production and patient's immune system.
  Cyclophosphamide: Alkylating agent which causes prevention of cell division by forming adducts with DNA Mesna: Medication used to decrease the risk of hemorrhagic cystitis rATG: lymphocyte-specific immunosuppressive agent Methylprednisolone: Steroid G-CSF: Granulocyte-colony stimulating factor; a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream Rituxan: Chimeric monoclonal antibody
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 23
Completed (Conditioning Regimen) | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] | 48.3 [27 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of Participants who Did Not Experience Treatment-Related Mortality
Time Frame: Mean 3.6 years
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 23
participants | 23

2. Secondary Outcome: Reduction of Muscle Relaxation Anti-spasmatic Medications
Description: Decrease (50%) and complete discontinuation of muscle relaxation anti-spasmatic medications
Time Frame: Mean 3.6 years
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 23
Participants | 14

3. Secondary Outcome: Short-form 36 Quality of Life Questionnaire (SF-36 QOL)
Description: Improvement is defined as a statistically significant change in SF-36 QOL score. The scale is 0-100. The lower the score the worse quality of life.
Time Frame: mean 3.6 years
Measure: Geometric Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 23
units on a scale
  Pre Treatment | 37.75 (12.81)
  Post Treatment | 58.35 (22.81)

ADVERSE EVENTS:
Time Frame: Up to 4.5 years
Arm/Group | Hematopoietic Stem Cell Transplantation
All-Cause Mortality (participants affected / at risk) | 1/23
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 5/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=23)
Non Treatment Related Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=23)
Hyperglycemia (Endocrine disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT02282514/Prot_SAP_000.pdf